CLINICAL TRIAL: NCT04706416
Title: N-Acetyl Glucosamine as Therapeutic Intervention for Coronavirus Disease-19 (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quantinosis.ai LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #2020-106
Record Dates: First submitted 2020-12-31; First posted 2021-01-12 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Coronavirus; Covid19
Keywords: N-acetyl glucosamine
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Acetylglucosamine

STUDY DESIGN:
Intervention Model Description: Patients with novel coronavirus (COVID-19) will be treated with N-acetylglucosamine (NAG) (700 mg every 12 hours) as first-line treatment for 30 days, along with standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-Acetyl Glucosamine (Experimental): All patients in the treatment arm of the study were treated with N-Acetyl Glucosamine, a potential therapy for Coronavirus Disease-19 (COVID-19).
  Interventions: Dietary Supplement: N-acetyl glucosamine (NAG)
- Control (Placebo Comparator): All patients in the comparator arm were admitted to the same hospital with COVID-19 but did not receive N-Acetyl Glucosamine treatment. All these patients were identified retrospectively.
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: N-acetyl glucosamine (NAG) — Patients with novel coronavirus (COVID-19) will be treated with N-acetylglucosamine (NAG) (700 mg every 12 hours) as first-line treatment for 30 days, along with standard of care.
  Arms: N-Acetyl Glucosamine
Other: Control — Patients do not receive treatment with N-Acetylglucosamine. They may receive other treatments at the discretion of the treating physician, as with the treatment group.
  Arms: Control

SUMMARY:
This study examines the efficacy of N-acetylglucosamine (NAG) in treating patients with novel coronavirus (COVID-19) infection.

DETAILED DESCRIPTION:
This is a single center, prospective, observational cohort study. A total of 150 cases who test positive for the novel coronavirus (COVID-19) will be recruited. Presenting to the emergency room of the study site, these cases will be treated with N-acetylglucosamine (NAG) in 700 mg doses every 12 hours as first-line treatment for 30 days. Standard of care (e.g., remdesivir approved for emergency use in severe cases, ventilator for patients with respiratory failure, etc.) will be provided based on the patient's clinical needs, which will be at the discretion of the treating physician. Upon admission, the research team will record patient demographics, comorbidities, symptoms, disease severity (as assessed by the World Health Organization Ordinal Scale for Clinical Improvement), need for supplemental oxygen, and time from symptom onset until hospital arrival. The research team will also collect bloodwork for the following at admission: white blood cell count (WBC), hematocrit (HCT), hemoglobin (HBG), C-reactive protein (CRP), procalcitonin (PCT), interleukin-6 (IL-6), and erythrocyte sedimentation rate (ESR). During the study period, discretionary treatments and interventions will be recorded daily until study exit. The primary outcomes of interest are rate of intubation, hospital length of stay, and mortality. Secondary outcomes of interest include intensive care unit (ICU) admission, ICU length of stay (LOS), supplemental oxygen duration, rate of hospice initiation, and poor clinical outcome (defined as combined death/hospice initiation).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Treated with N-acetyl glucosamine (NAG) as first-line treatment
* Present with coronavirus disease 2019 (COVID-19) symptoms (including but not limited to fever, cough, shortness of breath, sore throat, nasal congestion, malaise, headache, muscle pain, loss of taste and/or smell, diarrhea, and vomiting)
* Clinically diagnosed with COVID-19 by reverse transcription polymerase chain reaction (RT-PCR)
* No intubation prior to hospitalization and enrollment in the current study.

Exclusion Criteria:

* <18 years old upon admission
* Allergy to NAG
* Allergy to shellfish
* Currently taking warfarin
* Currently pregnant or lactating

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Valley Baptist Medical Center, Harlingen, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We will publish based on summary data, but make individual participant data available upon request. There are no plans to publish individual participant data.

REFERENCES:
- [Derived] Hassan AE. An observational cohort study to assess N-acetylglucosamine for COVID-19 treatment in the inpatient setting. Ann Med Surg (Lond). 2021 Aug;68:102574. doi: 10.1016/j.amsu.2021.102574. Epub 2021 Jul 16. PMID 34306677

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events in the study occurred after enrollment and prior to administration of the treatment.
Groups:
- N-Acetyl Glucosamine: All patients in the prospective arm of the study were treated with N-Acetyl Glucosamine, a potential therapy for Coronavirus Disease-19 (COVID-19).
  N-acetyl glucosamine (NAG): Patients with novel coronavirus (COVID-19) will be treated with N-acetylglucosamine (NAG) (700 mg every 12 hours) as first-line treatment for 30 days, along with standard of care.
- Control: All patients in the retrospective arm of the study were admitted to the same hospital for coronavirus disease 2019 (COVID-19), but they were not treated with the study treatment (N-Acetyl Glucosamine).
Period: Overall Study
Arm/Group | N-Acetyl Glucosamine | Control
Started | 50 | 100
Completed | 48 | 100
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: All patients in the comparative arm of the study were sampled retrospectively. All were admitted to the same hospital for coronavirus disease 2019 (COVID-19).
- Total: Total of all reporting groups
Arm/Group | N-Acetyl Glucosamine | Control | Total
Number analyzed (Participants) | 48 | 100 | 148
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [51.50 to 72.25] | 68 [57.25 to 76.75] | 67 [53.25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 38 | 62
  Male | 24 | 62 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 88 | 131
  Not Hispanic or Latino | 5 | 12 | 17
  Unknown or Not Reported | 0 | 0 | 0
Time from symptom onset [Median (Inter-Quartile Range); unit: days] | 12 [7 to 18.75] | 7 [4 to 15.75] | 8.5 [5 to 17]
Disease severity [Median (Inter-Quartile Range); unit: units on a scale] — World Health Organization (WHO) COVID-19 Disease Severity Score https://www.who.int/publications/i/item/WHO-2019-nCoV-clinical-2021-1
  One-time assessment at the time of hospital admission
  0 - not infected
  1. - mild illness (very few or mild symptoms)
  2. - mild illness (symptoms managed at home)
  3. - moderate illness (hospitalized, no supplemental oxygen)
  4. - moderate illness (hospitalized, supplemental oxygen)
  5. - severe illness (non-invasive breathing support)
  6. - severe illness (invasive breathing support)
  7. - severe illness (life-saving ventilation and organ support)
  8. - death
  units on a scale | 4 [4 to 5] | 4 [4 to 5] | 4 [4 to 5]
Supplemental oxygen use [Count of Participants; unit: Participants] | 46 | 86 | 132
White blood cell (WBC) [Median (Inter-Quartile Range); unit: x 10^9 cells/L] | 8.65 [6.05 to 11.73] | 10.25 [6.73 to 13.50] | 9.6 [6.33 to 13.2]
Hematocrit (hct) [Mean (Standard Deviation); unit: percentage of red blood cells] | 39.71 (6.02) | 37.97 (7.93) | 38.54 (7.385)
Hemoglobin (Hb) [Mean (Standard Deviation); unit: g/dL] | 12.69 (1.91) | 12.10 (2.61) | 12.3 (2.47)
Asthma [Count of Participants; unit: Participants] | 0 | 3 | 3
Atrial fibrillation [Count of Participants; unit: Participants] | 2 | 7 | 9
Coronary artery disease [Count of Participants; unit: Participants] | 6 | 17 | 23
Chronic heart failure [Count of Participants; unit: Participants] | 1 | 7 | 8
Chronic obstructive pulmonary disease (COPD) [Count of Participants; unit: Participants] | 3 | 11 | 14
End-stage renal disease (ESRD) [Count of Participants; unit: Participants] | 7 | 9 | 16
Hyperlipidemia [Count of Participants; unit: Participants] | 13 | 36 | 49
Hypertension [Count of Participants; unit: Participants] | 22 | 71 | 93
Obesity [Count of Participants; unit: Participants] | 27 | 40 | 67
Smoker [Count of Participants; unit: Participants] | 1 | 1 | 2
Positive chest x-ray [Count of Participants; unit: Participants] | 46 | 87 | 133
Received antibiotics [Count of Participants; unit: Participants] | 43 | 94 | 137
Received antivirals [Count of Participants; unit: Participants] | 13 | 6 | 19
Received corticosteroids [Count of Participants; unit: Participants] | 43 | 78 | 121
Received convalescent plasma [Count of Participants; unit: Participants] | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Intubated During Hospitalization
Description: The occurrence of intubation during hospitalization.
Time Frame: Through study completion (duration of patient's hospitalization), an average of 7-10 days.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetyl Glucosamine | Control
Number analyzed (Participants) | 48 | 100
Participants | 8 | 25
Statistical Analysis 1: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.297, Fisher Exact; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.26 to 1.48]
Statistical Analysis 2: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.541, Regression, Logistic; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.19 to 2.30]

2. Primary Outcome: Number of Participants Who Died During Hospitalization
Description: The occurrence of death during hospitalization.
Time Frame: Through study completion (duration of patient's hospitalization), an average of 7-10 days.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetyl Glucosamine | Control
Number analyzed (Participants) | 48 | 100
Participants | 6 | 28
Statistical Analysis 1: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.039, Fisher Exact; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.15 to 0.91]
Statistical Analysis 2: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.081, Regression, Logistic; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.09 to 1.07]

3. Primary Outcome: Hospital Length of Stay (LOS)
Description: The number of days the patient is hospitalized.
Time Frame: Through study completion (duration of patient's hospitalization), an average of 7-10 days and maximum of 30 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | N-Acetyl Glucosamine | Control
Number analyzed (Participants) | 48 | 100
days | 7 [5 to 11.75] | 7.5 [4 to 17]
Statistical Analysis 1: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.643, Wilcoxon (Mann-Whitney); Hodges-Lehmann estimator = 0, 95% CI 2-sided [-1.0 to 3.0]
Statistical Analysis 2: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.001, Regression, Linear; β-coefficient = -4.27, 95% CI 2-sided [-5.67 to -2.87]

4. Secondary Outcome: Number of Participants Admitted to Intensive Care Unit (ICU) During Hospitalization
Description: The occurrence of intensive care unit (ICU) admission.
Time Frame: Through study completion (duration of patient's hospitalization), an average of 7-10 days.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetyl Glucosamine | Control
Number analyzed (Participants) | 48 | 100
Participants | 11 | 36
Statistical Analysis 1: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.133, Fisher Exact; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.25 to 1.19]

5. Secondary Outcome: ICU Length of Stay
Description: The number of days the patient is in the ICU.
Time Frame: Through study completion (duration of patient's hospitalization), an average of 7-10 days and a maximum of 30 days.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- N-Acetyl Glucosamine: All patients in the treatment arm of the study were treated with N-Acetyl Glucosamine, a potential therapy for Coronavirus Disease-19 (COVID-19).
  10 treatment patients were admitted to the ICU and had ICU LOS data available.
- Control: All patients in the comparative arm of the study were sampled retrospectively. All were admitted to the same hospital for coronavirus disease 2019 (COVID-19).
  36 control patients were admitted to the ICU and had ICU LOS data available.
Arm/Group | N-Acetyl Glucosamine | Control
Number analyzed (Participants) | 11 | 36
days | 2.5 [0.75 to 14.75] | 9.0 [2.25 to 21.50]
Statistical Analysis 1: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.092, Wilcoxon (Mann-Whitney); Hodges-Lehmann estimator = 4.0, 95% CI 2-sided [-1.0 to 12.0]

6. Secondary Outcome: Supplemental Oxygen Duration
Description: The duration of supplemental oxygen use.
Time Frame: Through study completion (duration of patient's hospitalization), an average of 7-10 days and a maximum of 30 days.
Population: 46 treatment patients received supplemental oxygen support and had length of use data available. 86 control patients received supplemental oxygen support and had length of use data available.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | N-Acetyl Glucosamine | Control
Number analyzed (Participants) | 46 | 86
days | 7 [5 to 12] | 7 [3 to 15]
Statistical Analysis 1: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.834, Wilcoxon (Mann-Whitney); Hodges-Lehmann estimator = 0, 95% CI 2-sided [-2.0 to 2.0]

7. Secondary Outcome: Number of Participants Who Experienced Hospice Initiation During Hospitalization
Description: The occurrence of hospice proceedings initiation, indicating irreversible and imminent decline in health.
Time Frame: Through study completion (duration of patient's hospitalization), an average of 7-10 days.
Population: The hospice initiation cohort excludes those patients who died. 42 treatment patients survived and had hospice initiation data available. 72 control patients survived and had hospice initiation data available.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetyl Glucosamine | Control
Number analyzed (Participants) | 42 | 72
Participants | 0 | 4
Statistical Analysis 1: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.149, Fisher Exact; Odds Ratio (OR) = 0.001, 95% CI 2-sided [0 to 1.52]

8. Secondary Outcome: Number of Participants Who Experienced Poor Clinical Outcome During Hospitalization
Description: The occurrence of either death or initiation of hospice proceedings.
Time Frame: Through study completion (duration of patient's hospitalization), an average of 7-10 days.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetyl Glucosamine | Control
Number analyzed (Participants) | 48 | 100
Participants | 6 | 32
Statistical Analysis 1: Comparison: N-Acetyl Glucosamine vs Control; Test type: Superiority; p = 0.015, Fisher Exact; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.12 to 0.80]

ADVERSE EVENTS:
Time Frame: Patients were followed for the duration of the study period, which began at hospital admission/study enrollment and ended upon discharge, expiration, or 30 days.
Arm/Group | N-Acetyl Glucosamine | Control
All-Cause Mortality (participants affected / at risk) | 6/48 | 28/100
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/100
Other Adverse Events (participants affected / at risk) | 0/48 | 0/100

LIMITATIONS AND CAVEATS:
The conclusions that can be drawn from this study are limited by the relatively small number of participants, lack of randomization, use of a retrospective control arm, use of consecutive patients, temporality of different study arms in different stages of the pandemic, taking place at a single center, concomitant therapies, and potentially confounding baseline variables. These limitations were considered necessary costs in order to rapidly provide information during the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT04706416/Prot_SAP_000.pdf